CLINICAL TRIAL: NCT05136495
Title: Assessment of ADCY5-related Movement Disorders With Motion SENSors: a Feasibility Study
Brief Title: Assessment of ADCY5-related Movement Disorders With Motion SENSors
Acronym: SENSeo-ADCY5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: APHP201439; 2021-A00994-37 (Other: IDRCB Number)
Record Dates: First submitted 2021-04-29; First posted 2021-11-29 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: ADCY5-related Dyskinesia
Keywords: ADCY5; COFFEE; movement disorders
MeSH Terms: conditions — Dyskinesia, Familial, with Facial Myokymia; Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeinated coffee (Experimental): Drink caffeinated coffee one morning and drink decaffeinated coffee the other morning
  Interventions: Other: caffeinated coffee - decaffeinated coffee
- Decaffeinated coffee (Experimental): Drink decaffeinated coffee one morning and drink caffeinated coffee the other morning
  Interventions: Other: caffeinated coffee - decaffeinated coffee

INTERVENTIONS:
Other: caffeinated coffee - decaffeinated coffee — Drink caffeinated coffee one morning and drink decaffeinated coffee the other morning

SUMMARY:
ADCY5-related movement disorders are caused by dominant mutations in the ADCY5 gene. This rare neurogenetic disease is characterized by childhood-onset generalized hyperkinetic movements. Currently, the only tools available to rate the severity of movement disorders observed in ADCY5-patients are clinical rating scales of abnormal movements. These scales use the investigators' judgement to rate globally the severity of movements observed in various body parts of the patient. This protocol proposes to investigate a multimodal approach, combining a clinical scale assessment with ViconTM's objective movement measurement. A secondary objective of the study is to assess the effect of coffee on ADCY5-patients.

DETAILED DESCRIPTION:
ADCY5-related movement disorders are caused by dominant mutations in the ADCY5 gene. This rare neurogenetic disease is characterized by childhood-onset generalized hyperkinetic movements. The abnormal movements typically comprise a combination of dystonia, myoclonus and chorea occurring on a background of axial hypotonia, with superimposed disabling episodes of paroxysmal dyskinesia. The causing mutations are located in the ADCY5 gene coding for the Adenylate Cyclase 5 (AC5). AC5 is highly expressed in the striatal projection neurons of the striatum, a region involved in the control of movements. No effective treatment has been found. Currently, the only tools available to rate the severity of movement disorders observed in ADCY5-patients are clinical rating scales of abnormal movements. These scales use the investigators' judgement to globally rate movements severity in various body parts. This leads to inter-raters' scoring variability. An objective assessment through refined and comprehensive quantification of movements is needed. A motion capture system, such as ViconTM, could better reflect the global and focal variations of abnormal movements. This would be critical for the evaluation of responses to potential treatments. This protocol proposes to investigate a multimodal approach, combining a clinical scale assessment with ViconTM's objective movement measurement. A secondary objective of the study is to assess the effect of coffee on ADCY5-patients. The caffeine contained in coffee acts as a nonselective adenosine receptor antagonist, with a strong affinity for A2A receptors. By blocking A2A receptors, caffeine reduces the enzymatic activity of the altered mutated AC5 protein coded by the mutated ADCY5 gene. This effect could modulate the abnormal movements observed in patients.

ELIGIBILITY:
Inclusion Criteria:

* ADCY5 mutation carriers
* Age > 15 years old and 3 months
* Informed consent from the patient or/ and a legal representative when appropriate
* Affiliated with a social security system or beneficiary of such a regime or by waiver from CPP ( french ethic committee) for patients outside the European union ( EU)
* daily caffeine consumer

Exclusion Criteria:

* Hypersensitivity to caffeine or to xanthine derivatives
* Heart condition contraindicating coffee intake
* Liver failure
* Impaired comprehension interfering with an informed consent
* Positive pregnancy test for women of childbearing potential
* Patient treated by Enoxacin, Ciprofloxacin, Norfloxacin (Noroxin), Cimetidine, Phenytoin β-adrenergic drugs (β2 mimetics) at inclusion.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Quantification movement disorders | 24 HOURS
  Assessment of correlation between displacement data using the ViconTM system and standardized clinical scales' scores of movements

SECONDARY OUTCOMES:
Coffee effects | 24 Hours
  Change in abnormal movements, measured with motion sensors (ViconTM system) after caffeinated coffee vs after decaffeinated coffee
Involuntary scales evaluation | 24 Hours
  Change in abnormal movements, measured with standardized clinical scale (Abnormal Involuntary Movement Scale (AIMS; Global score range 0 to 28 and severity subscore range 0 to 4; higher scores mean worse outcome), after caffeinated coffee vs after decaffeinated coffee
Dyskinesia impairment evaluation | 24 Hours
  Change in abnormal movements, measured with standardized clinical scale Dyskinesia Impairment Scale (DIS) (total score range 0 to 288; higher scores mean worse outcome) after caffeinated coffee vs after decaffeinated coffee
Dyskinesia Rating Scale evaluation | 24 Hours
  Change in abnormal movements, measured with standardized clinical scale Unified Dyskinesia Rating Scale (UDysRS) (total score range of 0 to 104; higher scores mean worse outcome), after caffeinated coffee vs after decaffeinated coffee

CONTACTS AND LOCATIONS:
Locations (1):
- CIC Neurosciences, GH Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No